CLINICAL TRIAL: NCT02716246
Title: Phase I/II/III Gene Transfer Clinical Trial of scAAV9.U1a.hSGSH for Mucopolysaccharidosis (MPS) IIIA
Brief Title: Phase I/II/III Gene Transfer Clinical Trial of scAAV9.U1a.hSGSH
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABT-001; UX111-CL301 (Other: Ultragenyx Pharmaceutical Inc); 2015-003904-21 (EudraCT Number); 2023-510032-37-00 (EU CTIS Number)
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: MPS IIIA; Sanfilippo Syndrome; Sanfilippo A; Mucopolysaccharidosis III
Keywords: MPS IIIA; Sanfilippo; Gene Therapy
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Low Dose (Experimental): Dose of 0.5 X 10^13 vg/kg
  Interventions: Biological: UX111; Drug: Prophylactic Immunomodulatory (IM) Therapy; Drug: Adjuvant IM Therapy
- Cohort 2 Mid Dose (Experimental): Dose of 1 X 10^13 vg/kg
  Interventions: Biological: UX111; Drug: Prophylactic Immunomodulatory (IM) Therapy; Drug: Adjuvant IM Therapy
- Cohort 3 High Dose (Experimental): Dose of 3 X 10^13 vg/kg
  Interventions: Biological: UX111; Drug: Prophylactic Immunomodulatory (IM) Therapy; Drug: Adjuvant IM Therapy
- Cohort 4 High Dose (Spain Only) (Experimental): Dose of 3 X 10^13 vg/kg
  Interventions: Biological: UX111; Drug: Optimized Prophylactic IM Therapy; Drug: Adjuvant IM Therapy

INTERVENTIONS:
Biological: UX111 — Self-complementary adeno-associated virus serotype 9 carrying the human SGSH gene under the control of a U1a promoter (scAAV9.U1a.hSGSH) will be delivered one time through a venous catheter inserted into a peripheral limb vein.
  Other Names: scAAV9.U1a.hSGSH; ABO-102; rebisufligene etisparvovec
Drug: Prophylactic Immunomodulatory (IM) Therapy
  Arms: Cohort 1 Low Dose; Cohort 2 Mid Dose; Cohort 3 High Dose
Drug: Optimized Prophylactic IM Therapy
  Arms: Cohort 4 High Dose (Spain Only)
Drug: Adjuvant IM Therapy — The Principal Investigator and/or caregiver, in consultation with the medical monitor, will determine whether to initiate adjuvant IM therapy. Not all participants may receive adjuvant IM therapy.

SUMMARY:
The main objective of this study is to evaluate the efficacy and safety of UX111 for the treatment of MPS IIIA.

DETAILED DESCRIPTION:
Open-label, single dose, dose-escalation clinical trial of UX111 (scAAV9.U1a.hSGSH) injected intravenously through a peripheral limb vein. A limited course of prophylactic immunomodulatory (IM) therapy will be administered. At approved sites adjuvant IM therapy may be administered to selected participants. The Principal Investigator and/or caregiver, in consultation with the medical monitor, will determine whether to initiate adjuvant IM therapy. Not all participants may receive adjuvant IM therapy.

This study was previously posted by Abeona Therapeutics, Inc and was transferred to Ultragenyx in August 2022.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPS IIIA confirmed by the following methods:

  * No detectable or significantly reduced SGSH enzyme activity by leukocyte assay, and
  * Genomic DNA analysis demonstrating homozygous or compound heterozygous mutations in the SGSH gene (based upon review of documented results from a qualified laboratory, and with confirmation with Medical Monitor)
* Age:

  * For Cohort 1-3: From birth (participating sites in USA and Australia) OR 6 months (participating sites in Spain) to 2 years of age with no BSITD-III Cognitive Development Quotient (DQ) requirement, or older than 2 years with a BSITD-III Cognitive DQ of 60 or above (participating sites globally).
  * For Cohort 4 (participating sites in Spain): 3 months to ≤ 2 years of age with no BSITD-III Cognitive DQ requirement or > 2 years of age with a BSITD-III Cognitive DQ ≥ 60 (n = up to 6). Up to 2 additional subjects > 2 years and ≤ 5 years of age with a BSITD-III Cognitive DQ < 60 may also be enrolled. •Subjects must be ≥ 6 months of age before UX111 administration. However, subjects may be consented and initiate relevant Screening Procedures and IM treatment < 6 months of age. Refer to Section 8.2 for relevant screening procedures •For children ≤ 24 months chronological age who were born prematurely, defined as born at < 36 weeks gestational age, the corrected gestational age must be used for determining inclusion •The BSITD-III Cognitive DQ is assessed during the onsite Screening visit, for subjects who require it •The age of the child on the date of the Screening BSITD-III assessment is used to determine the requirement for the BSITD-III Cognitive DQ score.
* Cohort 4 only: Vaccination status based on age according to country-specific guidelines that is up to date 30 days prior to Enrollment as verified by documentation from the subject's primary care physician, and willing to defer vaccines through 6 months after completion of the subject's IM medication, or longer per Principal Investigator (PI) judgment. Emergency use authorization or conditional marketing authorization of coronavirus disease (COVID) vaccines is included unless there is an accepted medical exemption.

Exclusion Criteria:

* Inability to participate in the clinical evaluation as determined by PI
* Cohorts 1 to 3 only: Identification of two nonsense or null variants on genetic testing of the SGSH gene (based upon review of documented results from a qualified laboratory, and with confirmation with Medical Monitor)
* At least one S298P mutation in the SGSH gene (based upon review of documented results from a qualified laboratory, and with confirmation with Medical Monitor)
* Has evidence of an attenuated phenotype of MPS IIIA, in the judgement of the PI
* Presence of a concomitant medical condition that precludes lumbar puncture or use of anesthetics
* Active viral infection based on clinical observations
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer or precludes the child from participating in the protocol assessments and follow up
* Cohorts 1 to 3 only: Subjects with total anti-AAV9 antibody titers ≥ 1:100 equivalent to a positive screen as determined by ELISA binding assay in serum, Cohort 4 only: Subjects testing positive for total anti-AAV9 antibody titers in serum as determined at Screening
* Cohorts 1-3 only: Subjects with a positive response for the enzyme-linked immunosorbent spot assay (ELISpot) for T-cell responses to AAV9
* Cohorts 1-3 only: Serology consistent with exposure to human immunodeficiency virus (HIV), or serology consistent with active hepatitis B or C infection, Cohort 4: Current clinically significant infections (including any requiring systemic treatment including, but not limited to, HIV; hepatitis A, B, or C; varicella zosters virus; human T-cell lymphotropic virus type 1 [HTLV-1]; tuberculosis; or COVID-19) that would interfere with participation in the study.
* Bleeding disorder or any other medical condition or circumstance in which a lumbar puncture (for collection of CSF) is contraindicated according to local institutional policy
* Visual, hearing, or other impairment sufficient to preclude cooperation with neurodevelopmental testing
* Uncontrolled seizure disorder
* Any item (braces, etc.) or circumstance that would exclude the subject from being able to undergo MRI according to local institutional policy
* Any other situation that precludes the subject from undergoing procedures required in this study
* Subjects with cardiomyopathy or significant congenital heart abnormalities
* The presence of significant non-MPS IlIA related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
* Cohorts 1-3: Abnormal laboratory values Grade 2 or higher as defined in common terminology criteria for adverse events (CTCAE) v4.03 for gamma-glutamyl transferase (GGT), total bilirubin, creatinine, hemoglobin, white blood cell (WBC) count, platelet count, prothrombin time (PT) and activated partial thromboplastin time (aPTT), Cohort 4: Any of the following abnormal laboratory values from screening assessment:

  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), GGT, and/or alkaline phosphatase ≥ 2 × upper limit of normal (ULN) and/or total bilirubin > 1.5 × ULN
  * Anemia (hemoglobin < 10 g/dL)
  * Leukopenia or leukocytosis (total WBC count < 3,000/mm3 and > 15,000/mm3 respectively)
  * Abnormal absolute neutrophil count (ANC) of < 1000/mm3
  * Platelet count < 100,000/mm3
  * Coagulopathy (international normalized ratio [INR] > 1.5) or aPTT > 40 seconds
  * Renal impairment, defined as estimated glomerular filtration rate (eGFR) below the lower limit of normal (age and sex appropriate) based on Bedside Schwartz equation
* Female of childbearing potential who is pregnant or demonstrates a positive urine or bhCG result at screening assessment (if applicable)
* Cohorts 1-3: Any vaccination with viral attenuated vaccines less than 30 days prior to the scheduled date of treatment (and use of prednisolone)
* Previous treatment by hematopoietic stem cell transplantation
* Previous participation in a gene/cell therapy or enzyme replacement therapy (ERT) clinical trial

Cohort 4 only:

* Known hypersensitivity, that in the judgment of the PI, places the subject at increased risk for adverse effects.
* Unwilling to avoid consumption of grapefruit juice and the use of strong inhibitors of CYP3A4 and/or P-gp (eg, ketoconazole, voriconazole, itraconazole, erythromycin, telithromycin, or clarithromycin), strong inducers of CYP3A4 and/or P-gp (eg, rifampin, rifabutin, phenobarbital, carbamazepine, or phenytoin), and St. John's Wort from 30 days prior to Screening through completion of the IM regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-04-25 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Cerebrospinal Fluid (CSF) Heparan Sulfate (HS) (Disaccharide) Exposure | Up to Month 24 Visit
  Exposure is defined as the time-normalized area under the curve (AUC) of the percentage reduction from baseline.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development-Third Edition (BSITD-III) Cognitive Raw Score Over Time | Up to Month 24 Visit
CSF Ganglioside Type 2 (GM2) Exposure | Up to Month 24 Visit
  Exposure is defined as the time-normalized area under the curve (AUC) of the percentage change from baseline.
CSF Ganglioside Type 3 (GM3) Exposure | Up to Month 24 Visit
  Exposure is defined as the time-normalized area under the curve (AUC) of the percentage change from baseline.
Percent Change from Baseline in CSF HS | Baseline, Up to Month 24 Visit
BSITD-III Receptive Communication Raw Score Over Time | Up to Month 24 Visit
BSITD-III Expressive Communication Raw Score Over Time | Up to Month 24 Visit
Percent Change From Baseline in Total Cortical Volume | Baseline, Up to Month 24 Visit

OTHER OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events, and Treatment-Emergent Serious Adverse Events | Up to Month 24 Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (5):
- United States (2):
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Women's and Children's Hospital, North Adelaide, South Australia, Australia
- Spain (2):
  - Vall d'Hebron Barcelona Hospital Campus, Barcelona, Barcelona
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu H, Cataldi MP, Ware TA, Zaraspe K, Meadows AS, Murrey DA, McCarty DM. Functional correction of neurological and somatic disorders at later stages of disease in MPS IIIA mice by systemic scAAV9-hSGSH gene delivery. Mol Ther Methods Clin Dev. 2016 Jun 8;3:16036. doi: 10.1038/mtm.2016.36. eCollection 2016. PMID 27331076
- [Background] Fu H, Meadows AS, Pineda RJ, Kunkler KL, Truxal KV, McBride KL, Flanigan KM, McCarty DM. Differential Prevalence of Antibodies Against Adeno-Associated Virus in Healthy Children and Patients with Mucopolysaccharidosis III: Perspective for AAV-Mediated Gene Therapy. Hum Gene Ther Clin Dev. 2017 Dec;28(4):187-196. doi: 10.1089/humc.2017.109. Epub 2017 Oct 24. PMID 29064732
- [Derived] McCurdy VJ, Johnson AK, Gray-Edwards HL, Randle AN, Bradbury AM, Morrison NE, Hwang M, Baker HJ, Cox NR, Sena-Esteves M, Martin DR. Therapeutic benefit after intracranial gene therapy delivered during the symptomatic stage in a feline model of Sandhoff disease. Gene Ther. 2021 Apr;28(3-4):142-154. doi: 10.1038/s41434-020-00190-1. Epub 2020 Sep 3. PMID 32884151
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/